CLINICAL TRIAL: NCT01786317
Title: Measure of Ano-rectal Motility in Fecal Incontinence
Brief Title: Anal Motor Function in Fecal Incontinence
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/171/HP
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence, ano-rectal manometry
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fecal incontience: Patient with fecal incotinence who will be explored using high resoltuion manometry
  Interventions: Device: High resolution manometry
- Healthy controls: Healthy volunteers who will be explored using high resoltuion manometry
  Interventions: Device: High resolution manometry

INTERVENTIONS:
Device: High resolution manometry — Anorectal High resoltion manometry using electronic sensors

SUMMARY:
Traditionnal measurment of anorectal function is perfomed with manometric device using 2 to 3 pressure sensors. The investigators aim to evaluate the usefulness of high resolution manometry to measure anorectal motility

DETAILED DESCRIPTION:
Measurment of anorectal function is traditionnaly made using manometric device composed of perfused or ballon catheters. This allows the recording of anorectal pressure on 2-3 sites. Recently, high resolution manometryu devices using > 36 pressure channels have been developped. The investigators therefore aim to evaluate the usefullness of the high resolution manometry in patient with fecal incontinence in terms of feasability and diagnosis accuracy

ELIGIBILITY:
Inclusion Criteria:

* patient with fecal incontinence (group "fecal incontinence"
* subject without significant medical or surgical hisotry (group healthy controls)

Exclusion Criteria:

* pregnacy
* unable to speack/understand French language
* not affilitated to the French healthcare system
* history of anorectal disease (for the group of healthy controls) including fecal incontinence, or protocologic surgery
* constipation
* diarrhea

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heathy controls Patient with Fecal Incontience
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Anal squeezing pressure | Day 1
  measurement of anal squeezing pressure (mmhg)

SECONDARY OUTCOMES:
anal tone pressure | day 1
  measurement of anal tone pressure (mmhg)

CONTACTS AND LOCATIONS:
Overall Officials: guillaume Gourcerol, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, Normandy, France